CLINICAL TRIAL: NCT07070609
Title: Assessment of Sagittal Spine Balance in Patients Operated on for Anterior Chest Wall Funnel Deformity
Brief Title: Sagittal Spine Balance in Patients With Chest Wall Deformity
Status: Active, not recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: KB.006.134.2025
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Scoliosis Idiopathic Adolescent; Chest Deformities
Keywords: scoliosis; sagittal balance; anterior chest wall deformity
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sagittal balance disturbed

SUMMARY:
Does the funnel deformity affects the sagittal balance of the spine? This question is a result of a Principal Investigator's novel observation, that in some cases restoring the correct balance reduce the distance between the retracted sternum and the spine.

The aim of the study was to assess that sagittal balance of the spine change 6 months after surgical treatment?

We assess:

1. Deviations in sagittal balance in patients before the procedure by X-ray.
2. Change in the distance between the sternum and the anterior part of the nearest vertebral body after virtual reproduction of the correct sagittal balance by AI.
3. Change in the distance between the sternum and the anterior part of the nearest vertebral body 6 months after the Nuss procedure by X-ray.

DETAILED DESCRIPTION:
Assessment of sagittal spine balance in patients operated on for anterior chest wall funnel deformity.

Inclusion criteria:

age 10-18 idiopathic funnel chest Haller index above 3.2

Exclusion criteria:

Previous surgery within the chest and spine regions Anterior chest wall deformities caused by other disease syndromes (e.g. Marfan syndrome, Ehlers-Danlos syndrome) Haller index below 3.2

Study protocol:

1. Computed tomography of the chest.
2. Before the procedure, x-ray of the entire spine in a standing position, including the entire chest, pelvis and hip joints in the anterior and lateral projections (technical parameters will be provided separately).
3. Six months after the procedure, x-ray of the entire spine in a standing position, including the entire chest, pelvis and hip joints in the anterior and lateral projections (technical parameters will be provided separately).

The following are measured:

1. Haller index
2. Asymmetry index
3. Assessment of the Cobb angle in the case of disorders in the frontal plane - before and 6 months after the procedure
4. Assessment of the sagittal balance of the spine (details in a separate document) - before and 6 months after the procedure

We assess:

1. Deviations in sagittal balance in patients before the procedure by X-ray.
2. Change in the distance between the sternum and the anterior part of the nearest vertebral body after virtual reproduction of the correct sagittal balance by AI.
3. Change in the distance between the sternum and the anterior part of the nearest vertebral body 6 months after the Nuss procedure by X-ray.

Objective:

1. Does the funnel deformity affects the sagittal balance of the spine?
2. Does restoring the correct balance reduce the distance between the retracted sternum and the spine (AI)?
3. Does the sagittal balance of the spine change 6 months after surgical treatment?

ELIGIBILITY:
Inclusion Criteria:

* idiopathic funnel chest
* Haller index above 3.2

Exclusion Criteria:

* Previous surgery within the chest and spine regions
* Anterior chest wall deformities caused by other disease syndromes (e.g. Marfan syndrome, Ehlers-Danlos syndrome)
* Haller index below 3.2

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients operated on for anterior chest wall deformity.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
initial sagittal balance | 6 months
  Deviations in sagittal balance in patients before the procedure

SECONDARY OUTCOMES:
initial distance | 1 day
  Change in the distance between the sternum and the anterior part of the nearest vertebral body after virtual reproduction of the correct sagittal balance by AI.

OTHER OUTCOMES:
final sagittal balance | 6 months
  Change in the distance between the sternum and the anterior part of the nearest vertebral body 6 months after the Nuss procedure by X-ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Ortopedics Pomeranian Medical University,, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided
After asking of principal investigator